CLINICAL TRIAL: NCT01278173
Title: A Prospective, Open-label Study of the Structure and Function of the Retina in Adult Patients With Refractory Complex Partial Seizures Treated With Vigabatrin (Sabril®)
Brief Title: A Study of the Structure and Function of the Retina in Adult Patients With Refractory Complex Partial Seizures Treated With Vigabatrin (Sabril®)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Lundbeck LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 13098A
Record Dates: First submitted 2011-01-14; First posted 2011-01-17 (Estimated); Results first posted 2016-06-07 (Estimated); Last update posted 2016-06-07 (Estimated); Status verified 2016-04

CONDITIONS: Adult Refractory Complex Partial Seizures
Keywords: Vigabatrin-associated vision change; Adult refractory complex partial seizures; CPS; Epilepsy; Seizures; Brain diseases; Central Nervous System Diseases; Nervous System Diseases; Neurologic Manifestations; Enzyme Inhibitors; GABA Agents
MeSH Terms: conditions — Seizures; Epilepsy; Brain Diseases; Central Nervous System Diseases; Nervous System Diseases; Neurologic Manifestations | interventions — Vigabatrin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Sabril (Other)
  Interventions: Drug: Sabril

INTERVENTIONS:
Drug: Sabril — Sabril: 500 mg tablets, orally. Physicians will dose their patients according to guidance provided in the product label.
  Other Names: Vigabatrin

SUMMARY:
The purpose of the study is to evaluate the change in visual fields by means of automated static perimetry and to evaluate the change in retinal structure by means of spectral domain optical coherence tomography (SD-OCT) in adult patients with refractory complex partial seizures (CPS) being treated with vigabatrin (Sabril®)

DETAILED DESCRIPTION:
Multicenter, prospective open-label study with approximately 25 sites in the US that specialize in caring for adult patients with refractory CPS

* Sites must have access to Humphrey static perimetry and to Spectralis SD-OCT.
* All vision test results will be sent to the central readers for evaluation.
* Additional study tests:

  * The Columbia Suicide Severity Rating Scale (C-SSRS)
  * The National Eye Institute Visual Field Questionnaire-39 (NEI VFQ-39)
  * A whole blood sample for specific analysis of DNA characteristics
  * An optional whole blood sample for exploratory analysis of DNA characteristics
  * Plasma samples for bioanalytical analysis of vigabatrin and blood samples for taurine biomarker analysis

ELIGIBILITY:
Important Inclusion Criteria:

1. The patient speaks English or Spanish.
2. The patient has had no prior exposure to Sabril.
3. To begin Sabril therapy for the treatment of CPS.
4. Male or female ≥18 years of age.
5. The patient has refractory CPS:

   1. The patient has complex partial epilepsy of more than 1 year duration and no other seizure type within the past year except for partial seizures secondarily generalized.
   2. The patient has failed because of lack of efficacy 3 or more prior or concurrent treatment trials including 3 or more anti-epileptic drugs (AEDs) of differing pharmacologic mechanisms administered as monotherapy or polytherapy.
   3. The patient is taking at least 1 AED. A vagal nerve stimulator is not counted as an AED.
   4. The patient reports an average of 2 or more seizures per month averaged over the prior 3 months.
6. The patient is deemed by the treating neurologist and ophthalmologist to be able to reliably complete perimetry testing.
7. The initial (Visit 1) SD-OCT and static perimetry readings tests must be performed and assessed for technical adequacy by the SD-OCT and perimetry central readers prior to the first dose of Sabril. The initial (Visit 1) tangent corner test must be performed prior to the first dose of Sabril.

Exclusion Criteria:

1. Prior exposure to Sabril.
2. Pre-existing ocular or neurological disease that might affect bilateral visual fields or interfere with perimetry (e.g., aphakia, visually significant cataract, glaucoma, diabetes mellitus, ischemic optic neuropathy, multiple sclerosis). Patients with stable visual field defects from CNS lesions (e.g., epilepsy surgery more than 6 months prior to receiving Sabril) may be enrolled.
3. Concurrent exposure to medications with known or suspected retinal or optic nerve toxicity.
4. Concurrent use of an investigational agent or device or such use within 30 days of entering the study.
5. Concurrent use of the ketogenic or similar diet.
6. For any reason, the patient is considered by the investigator to be an unsuitable candidate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2010-12; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (22):
- United States (22):
  - California Pacific Medical Center, San Francisco, California
  - Yale Medical Center, New Haven, Connecticut
  - CNMRI, Dover, Delaware
  - Sunrise Clinical Research Group, Hollywood, Florida
  - University of South Florida, Tampa, Florida
  - Peachtree Neurological Clinic, Atlanta, Georgia
  - Idaho Comprehensive Epilepsy Center, Boise, Idaho
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - University of Kentucky Lexington, Lexington, Kentucky
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - Minnesota Epilepsy Group, PA, Saint Paul, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - Columbia University Medical Center, New York, New York
  - Neuroscience & Spine Institute, Charlotte, North Carolina
  - Oregon Health and Science University, Portland, Oregon
  - Thomas Jefferson University, Philadelphia, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Texas, Houston, Texas
  - Covenant Medical Group, Lubbock, Texas
  - University of Texas Health Science Center, San Antonio, Texas
  - Aurora BayCare Medical Center, Green Bay, Wisconsin
  - Aurora St. Luke's Medical Center, Milwaukee, Wisconsin

RESULTS

PARTICIPANT FLOW:
Groups:
- Sabril: Vigabatrin, 500 mg tablets, orally. Physicians will dose their patients according to guidance provided in the product label.
Period: Overall Study
Arm/Group | Sabril
Started | 65
Completed | 38
Not Completed | 27
Not completed — Lack of Efficacy | 13
Not completed — Adverse Event | 8
Not completed — Administrative or other reason | 4
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Population: All patients who took at least one dose of IMP.
Arm/Group | Sabril
Number analyzed (Participants) | 65
Age, Continuous [Mean (Standard Deviation); unit: years] | 39.8 (12.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 28
  Male | 37
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 2
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 58
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 65

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Reference Value in Field Width as Measured by 30-2 SITA Fast in Field Sensitivity (Mean Deviation - MD in dB)
Description: Mean change from the reference value in 30-2 SITA mean deviation, which was generated using the University of Iowa Visual Field Reading Center (VFRC) normative database and the Humphrey Field Analyzer (HFA) normative database. The reference value was defined as the average of the assessments performed at Visits 1 (baseline), 2 and 3 (first month of dosing). The mean change from the reference value are presented for Months 3, 6, 9 and 12. A negative change from the reference value indicates a decrease in the central visual field.
Time Frame: Baseline (Month 0), Month 3, Month 6, Month 9, Month 12
Population: All patients who had received at least one dose of investigational medicinal product and who had a valid reference value assessment and at least one valid post-reference value assessment. The total number of patients included in the analysis set was 55. The actual number of patients analysed for each time point and eye is presented below (N = x).
Measure: Mean (Standard Deviation); unit: dB
Arm/Group | Sabril
Number analyzed (Participants) | 55
dB
  VFRC database: Left eye, 3 months (N=50) | -0.28 (1.06)
  VFRC database: Left eye, 6 months (N=45) | -0.24 (1.13)
  VFRC database: Left eye, 9 months (N=39) | -0.14 (1.72)
  VFRC database: Left eye, 12 months (N=36) | -0.13 (1.58)
  VFRC database: Right eye, 3 months (N=50) | 0.08 (1.20)
  VFRC database: Right eye, 6 months (N=45) | -0.11 (1.40)
  VFRC database: Right eye, 9 months (N=39) | 0.02 (1.36)
  VFRC database: Right eye, 12 months (N=36) | -0.27 (1.61)
  HFA database: Left eye, 3 months (N=51) | -0.32 (1.13)
  HFA database: Left eye, 6 months (N=45) | -0.37 (1.15)
  HFA database: Left eye, 9 months (N=40) | -0.33 (1.61)
  HFA database: Left eye, 12 months (N=37) | -0.15 (1.68)
  HFA database: Right eye, 3 months (N=51) | 0.00 (1.18)
  HFA database: Right eye, 6 months (N=45) | -0.23 (1.40)
  HFA database: Right eye, 9 months (N=40) | -0.07 (1.33)
  HFA database: Right eye, 12 months (N=37) | -0.47 (1.60)

2. Primary Outcome: Change From Reference Value in Average RNFL (Retinal Nerve Fiber Layer) Thickness (µm) as Measured by SD-OCT (Spectral Domain-Optical Coherence Tomography)
Description: Mean change from the reference value in average RNFL thickness (µm) as measured by SD-OCT. The reference value was defined as the average of the assessments performed at Visits 1 (baseline), 2 and 3 (first month of dosing). Thinning of the RNFL, that is, a negative change from the reference value, has been associated with ophthalmological disease.
Time Frame: Baseline (Month 0), Month 3, Month 6, Month 9, Month 12
Population: All patients who had received at least one dose of IMP and who had a valid reference value assessment and at least one valid post-reference value assessment. The total number of patients included in the analysis set was 55. The actual number of patients analysed for each time point and eye is presented below (N = x).
Measure: Mean (Standard Deviation); unit: µm
Arm/Group | Sabril
Number analyzed (Participants) | 55
µm
  Left eye, 3 months (N=54) | 0.70 (2.56)
  Left eye, 6 months (N=48) | 4.15 (4.72)
  Left eye, 9 months (N=44) | 5.63 (4.30)
  Left eye, 12 months (N=39) | 6.45 (4.81)
  Right eye, 3 months (N=52) | 0.73 (2.20)
  Right eye, 6 months (N=47) | 4.21 (3.75)
  Right eye, 9 months (N=43) | 6.50 (4.67)
  Right eye, 12 months (N=39) | 7.19 (4.88)

ADVERSE EVENTS:
Time Frame: Baseline to end of study
Description: Treatment-Emergent Adverse Events are reported in this section
Arm/Group | Vigabatrin
Serious Adverse Events (participants affected / at risk) | 9/65
Other Adverse Events (participants affected / at risk) | 41/65
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Vigabatrin (N=65)
Atrial flutter (Cardiac disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Convulsion (Nervous system disorders) | 6
Partial seizures with secondary generalisation (Nervous system disorders) | 1
Postictal paralysis (Nervous system disorders) | 1
Postictal state (Nervous system disorders) | 1
Somnolence (Nervous system disorders) | 1
Suicidal ideation (Psychiatric disorders) | 1
Suicide attempt (Psychiatric disorders) | 1
Mitral valve repair (Surgical and medical procedures) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Vigabatrin (N=65)
Vision blurred (Eye disorders) | 6
Diarrhoea (Gastrointestinal disorders) | 4
Fatigue (General disorders) | 4
Fall (Injury, poisoning and procedural complications) | 8
Weight increased (Investigations) | 5
Convulsion (Nervous system disorders) | 13
Dizziness (Nervous system disorders) | 7
Somnolence (Nervous system disorders) | 4
Depression (Psychiatric disorders) | 4
Suicidal ideation (Psychiatric disorders) | 4
Vagal nerve stimulator implantation (Surgical and medical procedures) | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No